CLINICAL TRIAL: NCT00388531
Title: Multicenter, Prospective, Open Label Trial, Uncontrolled to Determine the Efficacy and Safety of Depocyt ® for the Treatment of CNS Relapse in Adult Patients With Lymphoblastic Leucemia or Very Aggressive Lymphoma
Brief Title: Depocyte in the Treatment of CNS Relapse in Patients With Lymphoblastic Leucemia or Very Aggressive Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-004414-17; DEPOCYLAN
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Lymphoblastic Leukemia; Lymphoma
Keywords: Acute Lymphoblastic Leucemia; Aggressive Non-Hodgkin-Lymphoma; CNS relapse; Cytarabine liposome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma

INTERVENTIONS:
Drug: Depocyte® — Depocyte® is a cytostatic drug

SUMMARY:
The first purpose is to confirm or not the efficacy of only one administration of DepoCyte®.

DETAILED DESCRIPTION:
It is a clinical study multicenter, prospective, open label trial, uncontrolled and nonrandomized

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphoblastic leukemia or very aggressive Non-Hodgkin-Lymphoma (Burkitt/Burkitt-like) and CNS relapse.

CNS involvement must be demonstrated by:

* A positive ventricular or lumbar CSF cytology defined as CSF cell counts > 5/µl (19/3 cells), obtained within 10 days prior to inclusion OR
* Characteristic signs and symptoms of neoplastic meningitis PLUS an MRI or CT scan indicating the presence of meningeal involvement. Patients with combined relapse in CNS and other locations may be included in case that systemic therapy with CNS active drugs (HDMTX;HDAC, Thiotepa) can be postponed for at least 2 weeks.
* Karnofsky >60%
* Age >18 years old
* Recovery from grade III/IV toxicities attributable to prior treatment with the exception of hematotoxicity.
* No severe heart, lung, liver or kidney dysfunction.
* The patient or guardian must be competent to provide informed consent and must provide written informed consent prior to the initiation of study procedures

Exclusion Criteria:

* Failure (as defined by no clearance of the CSF) to > 1 dose of prior intrathecal MTX or cytarabine or triple (MTX, ARAC, dexamethasone) therapy
* History of previous severe neurotoxicity (grade III-IV) attributed to intrathecal therapy or systemic high-dose therapy with methotrexate or cytarabine (vincristine induced peripheral neuropathy is accepted)
* Prior CNS relapse < 1 month before
* uncontrolled infection
* The patient must not be pregnant or breast feeding. If the patient is a female of child-bearing potential she must have a negative (urine or serum) pregnancy test and be using effective methods to prevent pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary purpose: | 1 year
response rate after one application of DepoCyte®. | 1 year

SECONDARY OUTCOMES:
Death in induction and in CR, Time to neurological progression, The frequency of improvement in pre-existing meningeal-disease related neurological symptoms,Karnofsky Performance Status,Survival,Toxicity according to CTCAE v.3 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Josep Mª Ribera, Doctor, Study Chair — Germans Trias i Pujol Hospital
Locations (9):
- Spain (9):
  - Hospital "Santa Creu i Sant Pau", Barcelona, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Salamanca, Salamanca

REFERENCES:
- [Background] Mastrangelo R, Poplack D, Bleyer A, Riccardi R, Sather H, D'Angio G. Report and recommendations of the Rome workshop concerning poor-prognosis acute lymphoblastic leukemia in children: biologic bases for staging, stratification, and treatment. Med Pediatr Oncol. 1986;14(3):191-4. doi: 10.1002/mpo.2950140317. No abstract available. PMID 3528788
- [Background] Gokbuget N, Hoelzer D. Meningeosis leukaemica in adult acute lymphoblastic leukaemia. J Neurooncol. 1998 Jun-Jul;38(2-3):167-80. doi: 10.1023/a:1005963732481. PMID 9696368
- [Background] Neale GA, Pui CH, Mahmoud HH, Mirro J Jr, Crist WM, Rivera GK, Goorha RM. Molecular evidence for minimal residual bone marrow disease in children with 'isolated' extra-medullary relapse of T-cell acute lymphoblastic leukemia. Leukemia. 1994 May;8(5):768-75. PMID 8182934
- [Background] Ribeiro RC, Rivera GK, Hudson M, Mulhern RK, Hancock ML, Kun L, Mahmoud H, Sandlund JT, Crist WM, Pui CH. An intensive re-treatment protocol for children with an isolated CNS relapse of acute lymphoblastic leukemia. J Clin Oncol. 1995 Feb;13(2):333-8. doi: 10.1200/JCO.1995.13.2.333. PMID 7844594
- [Background] Larson RA, Dodge RK, Burns CP, Lee EJ, Stone RM, Schulman P, Duggan D, Davey FR, Sobol RE, Frankel SR, et al. A five-drug remission induction regimen with intensive consolidation for adults with acute lymphoblastic leukemia: cancer and leukemia group B study 8811. Blood. 1995 Apr 15;85(8):2025-37. PMID 7718875
- [Background] Mandelli F, Annino L, Rotoli B. The GIMEMA ALL 0183 trial: analysis of 10-year follow-up. GIMEMA Cooperative Group, Italy. Br J Haematol. 1996 Mar;92(3):665-72. doi: 10.1046/j.1365-2141.1996.00394.x. PMID 8616033
- [Background] Morra E, Lazzarino M, Brusamolino E, Pagnucco G, Castagnola C, Bernasconi P, Orlandi E, Corso A, Santagostino A, Bernasconi C. The role of systemic high-dose cytarabine in the treatment of central nervous system leukemia. Clinical results in 46 patients. Cancer. 1993 Jul 15;72(2):439-45. doi: 10.1002/1097-0142(19930715)72:23.0.co;2-4. PMID 8319175
- [Background] Ellison RR, Mick R, Cuttner J, Schiffer CA, Silver RT, Henderson ES, Woliver T, Royston I, Davey FR, Glicksman AS, et al. The effects of postinduction intensification treatment with cytarabine and daunorubicin in adult acute lymphocytic leukemia: a prospective randomized clinical trial by Cancer and Leukemia Group B. J Clin Oncol. 1991 Nov;9(11):2002-15. doi: 10.1200/JCO.1991.9.11.2002. PMID 1941059
- [Background] Durrant IJ, Richards SM. Results of Medical Research Council trial UKALL IX in acute lymphoblastic leukaemia in adults: report from the Medical Research Council Working Party on Adult Leukaemia. Br J Haematol. 1993 Sep;85(1):84-92. doi: 10.1111/j.1365-2141.1993.tb08649.x. PMID 8251413
- [Background] Elonen E, Almqvist A, Hänninen A et al. Intensive treatment of acute lymphatic leukaemia in adults: ALL86 protocol. Haematologica. 1991;76 (Suppl 4):133
- [Background] Gökbuget N, Aguion-Freire E, Diedrich H et al. Characteristics and outcome of CNS relapse in patients with acute lymphoblastic leukemia (ALL) [abstract]. Blood. 1999;94:1287a.
- [Background] Gökbuget N, Arnold R, Eggeling B et al. Prospective evaluation of neurotoxicity of prophylactic intrathecal therapy in adult acute lymphoblastic leukemia. The Hematology Journal. 2000;1:591a.
- [Background] Chessells JM. Central nervous system directed therapy in acute lymphoblastic leukaemia. Baillieres Clin Haematol. 1994 Jun;7(2):349-63. doi: 10.1016/s0950-3536(05)80207-0. PMID 7803906
- [Background] Gagliano RG, Costanzi JJ. Paraplegia following intrathecal methotrexate: report of a case and review of the literature. Cancer. 1976 Apr;37(4):1663-8. doi: 10.1002/1097-0142(197604)37:43.0.co;2-7. PMID 946593
- [Background] Dunton SF, Nitschke R, Spruce WE, Bodensteiner J, Krous HF. Progressive ascending paralysis following administration of intrathecal and intravenous cytosine arabinoside. A Pediatric Oncology Group study. Cancer. 1986 Mar 15;57(6):1083-8. doi: 10.1002/1097-0142(19860315)57:63.0.co;2-b. PMID 3455842
- [Background] Bleyer WA, Poplack DG. Prophylaxis and treatment of leukemia in the central nervous system and other sanctuaries. Semin Oncol. 1985 Jun;12(2):131-48. No abstract available. PMID 3892694
- [Background] Glass JP, Lee YY, Bruner J, Fields WS. Treatment-related leukoencephalopathy. A study of three cases and literature review. Medicine (Baltimore). 1986 May;65(3):154-62. PMID 3517552
- [Background] Graham FL, Whitmore GF. The effect of-beta-D-arabinofuranosylcytosine on growth, viability, and DNA synthesis of mouse L-cells. Cancer Res. 1970 Nov;30(11):2627-35. No abstract available. PMID 5530557
- [Background] Zimm S, Collins JM, Curt GA, O'Neill D, Poplack DG. Cerebrospinal fluid pharmacokinetics of intraventricular and intravenous aziridinylbenzoquinone. Cancer Res. 1984 Apr;44(4):1698-701. PMID 6704975
- [Background] Murry DJ, Blaney SM. Clinical pharmacology of encapsulated sustained-release cytarabine. Ann Pharmacother. 2000 Oct;34(10):1173-8. doi: 10.1345/aph.19347. PMID 11054987
- [Background] Kim S, Chatelut E, Kim JC, Howell SB, Cates C, Kormanik PA, Chamberlain MC. Extended CSF cytarabine exposure following intrathecal administration of DTC 101. J Clin Oncol. 1993 Nov;11(11):2186-93. doi: 10.1200/JCO.1993.11.11.2186. PMID 8229133
- [Background] Chamberlain MC, Khatibi S, Kim JC, Howell SB, Chatelut E, Kim S. Treatment of leptomeningeal metastasis with intraventricular administration of depot cytarabine (DTC 101). A phase I study. Arch Neurol. 1993 Mar;50(3):261-4. doi: 10.1001/archneur.1993.00540030027009. PMID 8442704
- [Background] Chamberlain MC, Kormanik P, Howell SB, Kim S. Pharmacokinetics of intralumbar DTC-101 for the treatment of leptomeningeal metastases. Arch Neurol. 1995 Sep;52(9):912-7. doi: 10.1001/archneur.1995.00540330094020. PMID 7661730
- [Background] Glantz MJ, LaFollette S, Jaeckle KA, Shapiro W, Swinnen L, Rozental JR, Phuphanich S, Rogers LR, Gutheil JC, Batchelor T, Lyter D, Chamberlain M, Maria BL, Schiffer C, Bashir R, Thomas D, Cowens W, Howell SB. Randomized trial of a slow-release versus a standard formulation of cytarabine for the intrathecal treatment of lymphomatous meningitis. J Clin Oncol. 1999 Oct;17(10):3110-6. doi: 10.1200/JCO.1999.17.10.3110. PMID 10506606
- [Background] Howell SB. Liposomal cytarabine for the treatment of lymphomatous meningitis. Biological Therapy of Lymphoma. 2003;6:10-14.
- [Background] Glantz MJ, Jaeckle KA, Chamberlain MC, Phuphanich S, Recht L, Swinnen LJ, Maria B, LaFollette S, Schumann GB, Cole BF, Howell SB. A randomized controlled trial comparing intrathecal sustained-release cytarabine (DepoCyt) to intrathecal methotrexate in patients with neoplastic meningitis from solid tumors. Clin Cancer Res. 1999 Nov;5(11):3394-402. PMID 10589750
- [Background] Bomgaars J, Geyer J, Franklin J, et al. A phase I study of intrathecal liposomal cytarabine (DepoCyt) in pediatric patients with advanced meningeal malignancies. Proc Am Soc Clin Oncol. 2002;Abstract 433.
- [Background] Jaeckle KA, Phuphanich S, Bent MJ, Aiken R, Batchelor T, Campbell T, Fulton D, Gilbert M, Heros D, Rogers L, O'Day SJ, Akerley W, Allen J, Baidas S, Gertler SZ, Greenberg HS, LaFollette S, Lesser G, Mason W, Recht L, Wong E, Chamberlain MC, Cohn A, Glantz MJ, Gutheil JC, Maria B, Moots P, New P, Russell C, Shapiro W, Swinnen L, Howell SB. Intrathecal treatment of neoplastic meningitis due to breast cancer with a slow-release formulation of cytarabine. Br J Cancer. 2001 Jan;84(2):157-63. doi: 10.1054/bjoc.2000.1574. PMID 11161370
- [Background] Jaeckle KA, Batchelor T, O'Day SJ, Phuphanich S, New P, Lesser G, Cohn A, Gilbert M, Aiken R, Heros D, Rogers L, Wong E, Fulton D, Gutheil JC, Baidas S, Kennedy JM, Mason W, Moots P, Russell C, Swinnen LJ, Howell SB. An open label trial of sustained-release cytarabine (DepoCyt) for the intrathecal treatment of solid tumor neoplastic meningitis. J Neurooncol. 2002 May;57(3):231-9. doi: 10.1023/a:1015752331041. PMID 12125986
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- See also: Spanish association of Haematology — http://www.aehh.org
- See also: CRO — http://www.seif88.com